CLINICAL TRIAL: NCT00153205
Title: Serious Medication Errors in Pediatrics: Evaluation of Prevention Strategies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Patient Safety Foundation (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rainu Kaushal, MD, Rainu Kaushal, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005-P-000322/1; BWH
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Medication Errors
Keywords: medication errors; medical records systems, computerized; patient safety
MeSH Terms: interventions — Medical Order Entry Systems

ARMS (2):
- Introduction of A Clinical Pharmacist (Placebo Comparator)
  Interventions: Behavioral: computerized physician order entry
- Technological (Experimental)
  Interventions: Behavioral: computerized physician order entry

INTERVENTIONS:
Behavioral: computerized physician order entry

SUMMARY:
The purpose of this study is to determine how effective ward-based clinical pharmacists and computerized physician order entry systems are in reducing serious medication errors in pediatric inpatients.

DETAILED DESCRIPTION:
This is a prospective cohort study at Children's Hospital and Brigham and Women's Hospital (BWH), before and after the introduction of two distinct interventions. The first intervention at Children's Hospital was the introduction of clinical pharmacists on inpatient pediatric wards to target errors at the stages of physician ordering and nurse transcription. The second intervention is technological: the introduction of physician computer order entry at the BWH neonatal intensive care unit (NICU). This intervention will most effectively target errors at the stage of physician ordering, and secondarily address errors at the stage of pharmacy dispensing and nurse transcription. Data on serious medication errors will be collected pre and post each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the BWH NICU in the study pods during the study period

Exclusion Criteria:

* Patients in other units, non-study pods, or outside of the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-02; Primary Completion 2006-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
serious medication errors

CONTACTS AND LOCATIONS:
Overall Officials: Rainu Kaushal, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States